CLINICAL TRIAL: NCT02639676
Title: The Effects of Maternal Preeclampsia on the Development of Pulmonary and Vascular Dysfunction in Infants
Brief Title: Anti-Angiogenic Preeclampsia Milieu Impairs Infant Lung and Vascular Development
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Robert Tepper, MD, PhD, Indiana University
Other Study IDs: 1509123588; R01HL1222215 (Other Grant/Funding Number: National Heart, Lung, and Blood Institute)
Record Dates: First submitted 2015-12-10; First posted 2015-12-24 (Estimated); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Preeclampsia
Keywords: Infant; Bronchopulmonary Dysplasia; Premature
MeSH Terms: conditions — Pre-Eclampsia; Bronchopulmonary Dysplasia; Premature Birth | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Cord Blood, and Placenta Samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: Infants born to mothers with preeclampsia: Infants with expected delivery at 26+0 weeks gestation or greater .
  Interventions: Other: Diffusion Lung Capacity (DLCO), Vascular Challenge, Video Imaging, Specimen Collections
- Group 2: Infants born to mothers with normotensive pregnancies: Infants with expected delivery at 26+0 weeks gestation or greater.
  Interventions: Other: Diffusion Lung Capacity (DLCO), Vascular Challenge, Video Imaging, Specimen Collections

INTERVENTIONS:
Other: Diffusion Lung Capacity (DLCO), Vascular Challenge, Video Imaging, Specimen Collections

SUMMARY:
Pregnant mothers who develop high blood pressure and other vascular problems (preeclampsia) deliver babies with increased neonatal health problems, which include lung disease and vascular complications, later in life. Investigators will evaluate whether infants of mothers with preeclampsia have evidence for impaired development of the lungs and blood vessels.

DETAILED DESCRIPTION:
The overall objective of this study is to determine whether the anti-angiogenic environment of preeclampsia results in pulmonary and vascular dysfunction in infants. Specifically, study investigators hypothesize that the anti- angiogenic environment of preeclampsia will impair pulmonary development and promote vascular dysfunction in infants. Furthermore, study investigators hypothesize that circulating progenitor cell (CPC) measurements in cord blood will correlate with infant pulmonary (Aim #1) and systemic vascular (Aim #2) function. Study investigators will determine whether the pro-angiogenic circulating progenitor cells (CPC) versus non-circulating progenitor cells ratio in cord blood of pregnancies complicated by preeclampsia predicts pulmonary diffusing capacity and systemic vascular dysfunction, as well as respiratory distress syndrome (RDS) and bronchopulmonary dysplasia (BPD). This research represents an important translational study that extends observations made in pre-clinical animal models that have clearly established a critical relationship between angiogenesis and lung development. Preliminary data strongly suggest a relationship between pro-angiogenic circulating progenitor cells (CPCs), bronchopulmonary dysplasia (BPD), and pulmonary diffusion in human infants. Investigators will evaluate whether circulating progenitor cells (CPC)s are a biomarker for developing bronchopulmonary dysplasia (BPD), investigators will relate circulating progenitor cells (CPCs) to the underlying pathophysiology, as assessed by pulmonary function testing methods that we developed for this very difficult age group to evaluate. A positive finding in the study would provide the rationale for future translational studies evaluating the therapeutic potential of circulating progenitor cells (CPCs) to stimulate lung development of premature infants, as there are currently no known therapeutic interventions that minimize or prevent the development of bronchopulmonary dysplasia (BPD). One of several approaches could be applied in the future to increase circulating progenitor cells (CPCs) in premature infants: 1) pharmacologic mobilization of pro-angiogenic cells from the bone marrow, 2) expansion of pro-angiogenic cells from an infant's cord blood for autologous infusion, and 3) transfusion of pooled pro-angiogenic cells from multiple donors.

ELIGIBILITY:
Group 1: Infants born to mothers with preeclampsia

Inclusion Criteria:

* Clinical diagnosis of preeclampsia per the American College of Obstetricians and Gynecologists (ACOG) Task Force on Hypertension in Pregnancy 2013 report
* Anticipated delivery at 26+0 weeks gestation or greater.

Exclusion Criteria:

* Infant is not viable
* Cardiopulmonary defects
* Chest wall abnormalities
* Genetic anomalies
* Maternal history of Diabetes Mellitus
* Multiple gestation

Group 2: Infants born to mothers with normotensive pregnancies

Inclusion Criteria

* Normotensive pregnancy
* Anticipated delivery at 26+0 weeks gestation or greater.

Exclusion Criteria

* Maternal history of gestational diabetes
* Multiple gestation
* Genetic anomalies
* Chest wall abnormalities
* Chronic or Gestational hypertension
* Cardiopulmonary defects
* Infant is not viable

Min Age: 26 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Investigators are recruiting two groups of infants born at 26+0 weeks and greater. The first group are infant's born to mother's with preeclampsia and the second are infants born to mother's with a normotensive pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 292 (Actual)
Dates: Start 2016-02-11 (Actual); Primary Completion 2020-11-17 (Actual); Study Completion 2020-11-17 (Actual)

PRIMARY OUTCOMES:
Infant lung development measured by diffusion lung capacity (DLCO) | by month 8

SECONDARY OUTCOMES:
Airway function measured by spirometry | by month 8

OTHER OUTCOMES:
Lung development measured by angiogenic growth factors: ratio of circulating progenitor cells to non circulating progenitor cells, vascular endothelial growth factor, and soluble fms-like tyrosine kinase-1 found in cord blood. | by month 8
Systemic vascular function measured by angiogenic factors of the ratio of circulating progenitor cells to non progenitor cells, vascular endothelial growth factor, and soluble fms-like tyronsine kinase-1 found in cord blood. | by month 8
Systemic vascular function measured by a vascular challenge on capillary density. | by month 8
Systemic vascular function measured by blood pressure. | by month 8

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Tepper, MD, PhD, Principal Investigator — Indiana University
Locations (1):
- Riley Hospital for Children, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided